CLINICAL TRIAL: NCT04746079
Title: Positive Imagery Therapy and the Incidence of Emergence Reactions With the Use of Ketamine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mercy Health Ohio (Other)
Collaborators: Lake Erie College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-025
Record Dates: First submitted 2021-02-08; First posted 2021-02-09 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-05

CONDITIONS: Procedural Sedation; Emergence Delirium
Keywords: ketamine
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: The sealed envelope method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Imagery Therapy (Experimental): Perform procedural sedation with slow push of ketamine, 1.5mg/kg, over thirty seconds while reading the Positive Imagery Therapy below:
  "Relax and close your eyes. Take deep breaths in through your nose and out through your mouth as you listen to the sound of my voice. (Three second pause.) I want you to picture yourself lying on a towel on a soft sandy beach. (Three second pause.) You can see a palm trees swaying in the wind beneath a bright blue sky with a few white puffy clouds. (Three second pause.) You can feel the sand between your toes, the warm sunlight on your skin and a cool breeze. (Three second pause) You can smell coconut lotion in the breeze. (Three second pause.) You can hear the sound of waves gently crashing on the beach and seagulls crying in the distance. **End of vignette**
  Interventions: Behavioral: Positive Imagery Therapy
- Control (No Intervention): Perform procedural sedation with slow push of ketamine, 1.5mg/kg, over thirty seconds with no positive imagery therapy.

INTERVENTIONS:
Behavioral: Positive Imagery Therapy — Perform procedural sedation with slow push of ketamine, 1.5mg/kg, over thirty seconds while reading the Positive Imagery Therapy.
  Arms: Positive Imagery Therapy

SUMMARY:
The purpose of this study is to determine if positive imagery therapy while using ketamine in procedural sedation reduces the number of emergence reactions and impacts pre and post-procedural anxiety.

DETAILED DESCRIPTION:
This is a multi-center, randomized controlled trial looking at if positive imagery therapy while using ketamine during procedural sedation will reduce the number of emergence reactions and impacts pre and post procedural anxiety. After informed consent has been established and the subject is determined to meet eligibility criteria, participants will be randomized into 2 groups. The interventional group will undergo positive imagery therapy during sedation and the control will not. The duration of subject participation will be from the onset of sedation beginning until the patient is recovered.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* requires procedural sedation in the emergency department for whom ketamine is selected by the provider as the medication for procedural sedation

Exclusion Criteria:

* age below 18 years of age
* any patient with a contraindication to the use of ketamine for the procedural sedation
* any prisoners
* pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Richmond Agitation Sedation Score (RASS) for those receiving procedural sedation with and without ketamine | From beginning of ketamine administration until patient returns to baseline. Estimated less than 1 hour.
  RASS score measured is -5 to +4. A lower score indicates someone is more alert, calm, drowsy indicating the patient has no emergence reaction. Higher score indicates an emergence reaction occurred.
Pittsburgh Agitation Score for those receiving procedural sedation with and without ketamine | From beginning of ketamine administration until patient returns to baseline. Estimated less than 1 hour.
  PAS is measures from 0-16. A lower score indicated no agitation or emergence reaction while a higher score does.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bolotin, MD, Principal Investigator — Bon Secours Mercy Health
Locations (1):
- Mercy Health St Elizabeth Youngstown, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sener S, Eken C, Schultz CH, Serinken M, Ozsarac M. Ketamine with and without midazolam for emergency department sedation in adults: a randomized controlled trial. Ann Emerg Med. 2011 Feb;57(2):109-114.e2. doi: 10.1016/j.annemergmed.2010.09.010. PMID 20970888
- [Background] Akhlaghi N, Payandemehr P, Yaseri M, Akhlaghi AA, Abdolrazaghnejad A. Premedication With Midazolam or Haloperidol to Prevent Recovery Agitation in Adults Undergoing Procedural Sedation With Ketamine: A Randomized Double-Blind Clinical Trial. Ann Emerg Med. 2019 May;73(5):462-469. doi: 10.1016/j.annemergmed.2018.11.016. Epub 2019 Jan 3. PMID 30611640
- [Background] Stoker AD, Rosenfeld DM, Buras MR, Alvord JM, Gorlin AW. Evaluation of Clinical Factors Associated with Adverse Drug Events in Patients Receiving Sub-Anesthetic Ketamine Infusions. J Pain Res. 2019 Dec 23;12:3413-3421. doi: 10.2147/JPR.S217005. eCollection 2019. PMID 31920366
- [Background] Schwenk ES, Goldberg SF, Patel RD, Zhou J, Adams DR, Baratta JL, Viscusi ER, Epstein RH. Adverse Drug Effects and Preoperative Medication Factors Related to Perioperative Low-Dose Ketamine Infusions. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):482-7. doi: 10.1097/AAP.0000000000000416. PMID 27281730
- [Background] Sherwin TS, Green SM, Khan A, Chapman DS, Dannenberg B. Does adjunctive midazolam reduce recovery agitation after ketamine sedation for pediatric procedures? A randomized, double-blind, placebo-controlled trial. Ann Emerg Med. 2000 Mar;35(3):229-38. doi: 10.1016/s0196-0644(00)70073-4. PMID 10692189
- [Background] Vardy JM, Dignon N, Mukherjee N, Sami DM, Balachandran G, Taylor S. Audit of the safety and effectiveness of ketamine for procedural sedation in the emergency department. Emerg Med J. 2008 Sep;25(9):579-82. doi: 10.1136/emj.2007.056200. PMID 18723707
- [Background] Newton A, Fitton L. Intravenous ketamine for adult procedural sedation in the emergency department: a prospective cohort study. Emerg Med J. 2008 Aug;25(8):498-501. doi: 10.1136/emj.2007.053421. PMID 18660398
- [Background] Strayer RJ, Nelson LS. Adverse events associated with ketamine for procedural sedation in adults. Am J Emerg Med. 2008 Nov;26(9):985-1028. doi: 10.1016/j.ajem.2007.12.005. PMID 19091264
- [Background] Green SM, Roback MG, Krauss B, Brown L, McGlone RG, Agrawal D, McKee M, Weiss M, Pitetti RD, Hostetler MA, Wathen JE, Treston G, Garcia Pena BM, Gerber AC, Losek JD; Emergency Department Ketamine Meta-Analysis Study Group. Predictors of emesis and recovery agitation with emergency department ketamine sedation: an individual-patient data meta-analysis of 8,282 children. Ann Emerg Med. 2009 Aug;54(2):171-80.e1-4. doi: 10.1016/j.annemergmed.2009.04.004. Epub 2009 Jun 6. PMID 19501426
- [Background] Treston G, Bell A, Cardwell R, Fincher G, Chand D, Cashion G. What is the nature of the emergence phenomenon when using intravenous or intramuscular ketamine for paediatric procedural sedation? Emerg Med Australas. 2009 Aug;21(4):315-22. doi: 10.1111/j.1742-6723.2009.01203.x. PMID 19682018
- [Background] Somashekara SC, Govindadas D, Devashankaraiah G, Mahato R, Deepalaxmi S, Srinivas V, Murugesh JV, Devanand. Midazolam premedication in attenuating ketamine psychic sequelae. J Basic Clin Pharm. 2010 Sep;1(4):209-13. Epub 2010 Nov 15. PMID 24825990
- [Background] Trivedi S, Kumar R, Tripathi AK, Mehta RK. A Comparative Study of Dexmedetomidine and Midazolam in Reducing Delirium Caused by Ketamine. J Clin Diagn Res. 2016 Aug;10(8):UC01-4. doi: 10.7860/JCDR/2016/18397.8225. Epub 2016 Aug 1. PMID 27656531
- [Background] Perumal DK, Adhimoolam M, Selvaraj N, Lazarus SP, Mohammed MA. Midazolam premedication for Ketamine-induced emergence phenomenon: A prospective observational study. J Res Pharm Pract. 2015 Apr-Jun;4(2):89-93. doi: 10.4103/2279-042X.155758. PMID 25984547
- [Background] Bergman SA. Ketamine: review of its pharmacology and its use in pediatric anesthesia. Anesth Prog. 1999 Winter;46(1):10-20. PMID 10551055
- [Background] Roback MG, Wathen JE, Bajaj L, Bothner JP. Adverse events associated with procedural sedation and analgesia in a pediatric emergency department: a comparison of common parenteral drugs. Acad Emerg Med. 2005 Jun;12(6):508-13. doi: 10.1197/j.aem.2004.12.009. PMID 15930401
- [Background] Cheong SH, Lee KM, Lim SH, Cho KR, Kim MH, Ko MJ, Shim JC, Oh MK, Kim YH, Lee SE. Brief report: the effect of suggestion on unpleasant dreams induced by ketamine administration. Anesth Analg. 2011 May;112(5):1082-5. doi: 10.1213/ANE.0b013e31820eeb0e. Epub 2011 Feb 23. PMID 21346162
- [Background] Asl Aminabadi N, Erfanparast L, Sohrabi A, Ghertasi Oskouei S, Naghili A. The Impact of Virtual Reality Distraction on Pain and Anxiety during Dental Treatment in 4-6 Year-Old Children: a Randomized Controlled Clinical Trial. J Dent Res Dent Clin Dent Prospects. 2012 Fall;6(4):117-24. doi: 10.5681/joddd.2012.025. Epub 2012 Nov 12. PMID 23277857
- [Background] Huet A, Lucas-Polomeni MM, Robert JC, Sixou JL, Wodey E. Hypnosis and dental anesthesia in children: a prospective controlled study. Int J Clin Exp Hypn. 2011 Oct-Dec;59(4):424-40. doi: 10.1080/00207144.2011.594740. PMID 21867378
- [Background] Heilbrunn BR, Wittern RE, Lee JB, Pham PK, Hamilton AH, Nager AL. Reducing anxiety in the pediatric emergency department: a comparative trial. J Emerg Med. 2014 Dec;47(6):623-31. doi: 10.1016/j.jemermed.2014.06.052. Epub 2014 Sep 27. PMID 25271180